CLINICAL TRIAL: NCT00216866
Title: A Pilot Study of Central Venous Catheter Survival in Cancer Patients Using Low Molecular Weight Heparin (Dalteparin) for the Treatment of Deep Vein Thrombosis of the Upper Extremity
Brief Title: The Catheter Study: Central Venous Catheter Survival in Cancer Patients Using Low Molecular Weight Heparin (Dalteparin) for the Treatment of Deep Vein Thrombosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-02-191
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Embolism and Thrombosis
Keywords: Embolism; Thrombosis
MeSH Terms: conditions — Embolism and Thrombosis; Embolism; Thrombosis | interventions — Dalteparin; Warfarin

INTERVENTIONS:
Drug: Dalteparin
Drug: Warfarin

SUMMARY:
The purpose of this study is to obtain an estimate of catheter survival in the setting of upper extremity deep vein thrombosis (UEDVT) in patients treated with dalteparin and warfarin.

Anticoagulation with dalteparin and warfarin in patients with UEDVT secondary to central venous catheters in patients with an active malignancy is an effective therapy as quantified by the success of catheter preservation. A prolonged line salvage rate without a recurrence of UEDVT will improve the management of cancer patients who develop upper extremity deep venous thrombosis in the setting of a central venous (CV) catheter.

DETAILED DESCRIPTION:
Deep venous thrombosis (DVT) is a serious disorder with an annual incidence of approximately 0.1% and increasing with age to 1% in the elderly. Deep venous thrombosis of the upper extremity (UEDVT) is estimated to constitute 1-5% of all cases of DVT.

The therapy of UEDVT has not been standardized.Therapeutic options include anticoagulation with unfractionated heparin followed by warfarin, treatment with a thrombolytic agent, or a thrombectomy. Recently, treatment with low molecular weight heparin has been shown to be a safe and effective treatment for patients with verified UEDVT.

In patients with cancer, treatment of UEDVT associated with central venous catheters is even less standardized. Some groups advocate removal of the catheter as the sole treatment for the DVT, others remove the catheter and treat the DVT. A major disadvantage to removing the line is that often re-insertion in the opposite limb is then required to avoid disruption of chemotherapeutic treatment. This reinsertion again puts the patient at risk for thrombosis and pulmonary embolism. Another therapy is treatment only with systemic thrombolytic therapy. The disadvantage of thrombolytic therapy in persons with cancer is that there is a high risk for major bleeding at the doses used.

A treatment regimen that has been adopted by the London Health Sciences Centre, and others across Canada, is to leave the catheter in place and treat the DVT with low molecular weight heparin and warfarin. This regimen is believed to halt the progression of thrombi, prevent embolism and allow natural thrombolytic mechanisms to work effectively. By leaving the central line in situ and appropriately treating the thrombosis there is no disruption in the delivery of life-prolonging or life-saving treatment in the form of chemotherapy.

Preliminary data has been collected over the past 24 months at the London Health Sciences Centre; the results suggest that this approach to treatment will prove to be beneficial to the patient. Thirteen (13) patients with cancer and an UEDVT associated with a central venous catheter were treated with dalteparin and warfarin with an intention to leave the central line in situ. Of the 13, 1 patient had the line removed after 3 days at a peripheral hospital against recommendation. The UEDVT was treated successfully and without the need for line removal in 9 (75%) of the remaining 12 patients. Two (2) of the 12 had lines removed at 1 week and 1 had the line removed at 4 weeks due to worsening symptoms of UEDVT.

Therefore, UEDVT is a more common and less benign disease than previously reported and generally arises in the presence of recognizable risk factors such as central venous catheters and cancer. Treatment of the UEDVT with dalteparin and warfarin will treat the thrombosis while preserving the central venous access for continued use. Hence, the need for additional catheters and subsequent risk of bilateral UEDVT will be minimized.

Result of the CLOT (Clot in Cancer) Trial have shown the superiority of treatment with dalteparin for 6 months as compared to the conventional treatment with short-term dalteparin and extended warfarin for cancer patients with acute symptomatic DVT or PE. Extended anticoagulant therapy may be beneficial in patients with UEDVT as well, however, there are currently no estimates of clinical outcomes for either conventional (dalteparin followed by warfarin) or extended therapy with dalteparin in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Males or females greater than or equal to 18 years of age, inclusive.
* Symptomatic acute upper limb thrombosis with or without pulmonary embolism associated with central venous catheter objectively documented by compression ultrasonography, venogram or computed tomography (CT) scan.
* Diagnosis of active malignancy, as defined by patients who are either receiving active treatment, or have metastatic disease or who have been diagnosed within the past two years.
* Willing to provide written informed consent.

Exclusion Criteria:

* Dialysis catheters.
* Active bleeding or high risk for major bleeding.
* Platelet count < 100 x 10x9/L.
* Serum creatinine > 177umol/L
* Currently on warfarin with therapeutic intent (does not include minidose warfarin used as prophylaxis for CV catheter thrombosis).
* Pulmonary embolism accompanied by hemodynamic instability or oxygen requirement.
* Inability to infuse through the catheter after a trial of intraluminal thrombolytic therapy.
* Patients with acute myelogenous leukemia (AML) or acute lymphoblastic leukemia (ALL) with a bone marrow or stem cell transplant pending in next 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2002-09 (Actual); Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study will be rate of central line failure, defined as infusion failure that does not respond to 2mg tissue plasminogen activator (tPA), within the 3 months of study follow-up.

SECONDARY OUTCOMES:
The secondary endpoints include recurrence of deep vein thrombosis (DVT) or pulmonary embolism (PE), major bleeding and death, time to central line failure.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Kovacs, MD, FRCPC, Principal Investigator — The University of Western Ontario
Locations (6):
- Canada (6):
  - Queen Elizabeth II Health Care Centre, Halifax, Nova Scotia
  - St. Joseph's Healthcare, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa General Hospital, Ottawa, Ontario
  - Ottawa Civic Hospital, Ottawa, Ontario
  - Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Background] Kommareddy A, Zaroukian MH, Hassouna HI. Upper extremity deep venous thrombosis. Semin Thromb Hemost. 2002 Feb;28(1):89-99. doi: 10.1055/s-2002-20567. PMID 11885029
- [Background] Kooij JD, van der Zant FM, van Beek EJ, Reekers JA. Pulmonary embolism in deep venous thrombosis of the upper extremity: more often in catheter-related thrombosis. Neth J Med. 1997 Jun;50(6):238-42. doi: 10.1016/s0300-2977(97)00020-x. PMID 9232088
- [Background] Monreal M, Raventos A, Lerma R, Ruiz J, Lafoz E, Alastrue A, Llamazares JF. Pulmonary embolism in patients with upper extremity DVT associated to venous central lines--a prospective study. Thromb Haemost. 1994 Oct;72(4):548-50. PMID 7878630
- [Background] Volturo GA, Repeta RJ Jr. Non-lower extremity deep vein thrombosis. Emerg Med Clin North Am. 2001 Nov;19(4):877-93, vi. doi: 10.1016/s0733-8627(05)70224-8. PMID 11762277
- [Background] Monreal M, Davant E. Thrombotic complications of central venous catheters in cancer patients. Acta Haematol. 2001;106(1-2):69-72. doi: 10.1159/000046591. PMID 11549779
- [Background] Elliott G. Upper-extremity deep vein thrombosis. Lancet. 1997 Apr 26;349(9060):1188-9. doi: 10.1016/S0140-6736(05)62408-7. No abstract available. PMID 9130936
- [Background] Baarslag HJ, van Beek EJ, Koopman MM, Reekers JA. Prospective study of color duplex ultrasonography compared with contrast venography in patients suspected of having deep venous thrombosis of the upper extremities. Ann Intern Med. 2002 Jun 18;136(12):865-72. doi: 10.7326/0003-4819-136-12-200206180-00007. PMID 12069560
- [Background] Savage KJ, Wells PS, Schulz V, Goudie D, Morrow B, Cruickshank M, Kovacs MJ. Outpatient use of low molecular weight heparin (Dalteparin) for the treatment of deep vein thrombosis of the upper extremity. Thromb Haemost. 1999 Sep;82(3):1008-10. PMID 10494754
- [Background] Kovacs MJ, Anderson DA, Wells PS. Prospective assessment of a nomogram for the initiation of oral anticoagulation therapy for outpatient treatment of venous thromboembolism. Pathophysiol Haemost Thromb. 2002 May-Jun;32(3):131-3. doi: 10.1159/000065215. PMID 12372927